CLINICAL TRIAL: NCT02029014
Title: Evaluation of Safety and Efficacy of the New Generation of Left Appendage Closure With the LAmbre Device in AF Patients Not Suitable for Use of Warfarin
Brief Title: Safety and Efficacy Study of LAmbre LAA Closure Device for Treating AF Patients Who Cannot Take Warfarin
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lifetech Scientific (Shenzhen) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LAA v1.1
Record Dates: First submitted 2014-01-06; First posted 2014-01-07 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Atrial Fibrillation
Keywords: LAmbre
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LAmbre closure system (Experimental)
  Interventions: Device: LAA closure system

INTERVENTIONS:
Device: LAA closure system

SUMMARY:
The aim of this study is to assess the efficacy, safety and performance of LAmbre left atrial appendage closure system in patients with non-valvular atrial fibrillation who cannot be treated with Warfarin.

ELIGIBILITY:
Inclusion Criteria:

* Age>=18, CHADS2 score>=1
* Patients cannot be treated long-term with Warfarin
* Eligible for clopidogrel and aspirin
* Provide written informed consent and agree to comply with required follow-ups

Exclusion Criteria:

* Need to take Warfarin
* Presence of rheumatic, degenerative or congenital valvular heart diseases
* Early stage or paroxysmal AF
* Symptomatic patients with carotid artery disease (such as carotid stenosis>=50%)
* Heart failure NYHA grade IV
* Recent 30 days stroke or TIA
* Presence of active sepsis or endocarditis
* Cardiac tumors or other malignancy with estimated life expectancy <2 years
* Abnormal blood test; renal disfunction
* LAA removed or heart implant patients
* Patients have planned electrophysiological ablation or cardioversion 30 days post implantation of the LAmbre system
* Patients have history of mechanical prosthesis operation
* Patients who are pregnant, or desire to be pregnant during the during the study
* Participation in other trials
* A known allergy to nitinol
* Patients will not be able to complete the trial

Esophageal ultrasonic exclusion criteria:

* LAA Ostium <=12mm or >=30mm
* LVEF <30%
* Presence of thrombus in the heart
* High risk PFO
* Mitral valve stenosis (valve area <2 cm2

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2014-03; Primary Completion 2016-03 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Ischemic stroke | One year
Successful sealing of the LAA | One year

SECONDARY OUTCOMES:
Component events | One year
  death, thromboembolism, device related complication and MACCE
MACCE | One year
  all-cause death, stroke, cardiac tamponade and renal failure
Complication at puncture site | One year
Device performance assessed by TEE/TTE | One year
  Device migration/embolization Regurgitation Perivalvular leak

CONTACTS AND LOCATIONS:
Overall Officials: Congxin Huang, MD, Principal Investigator — People's Hospital of Wuhan University
Locations (1):
- People's Hospital of Wuhan University, Wuhan, Hubei, China